CLINICAL TRIAL: NCT05045872
Title: Clinical Study of Domestic Polysaccharide Superparamagnetic Iron Oxide Nanoparticle Injection for Renal Contrast-enhanced Magnetic Resonance Imaging
Brief Title: Assessment of Renal Vasculature and Function with Ferumoxytol-enhanced Magnetic Resonance Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 013
Record Dates: First submitted 2021-08-21; First posted 2021-09-16 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Ultrasmall Superparamagnetic Particles of Iron Oxide; Contrast-Enhanced Magnetic Resonance; Renal Artery Stenosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Artery Obstruction | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ferumoxytol-enhanced renal magnetic resonance imaging (Experimental): Patients will receive ferumoxytol-enhanced renal magnetic resonance imaging before renal angiography. Ferumoxytol (510 mg/17mL; Chia Tai Tianqing Pharmaceutical Group Co Ltd, Nanjing, China) will be diluted at 1:4 (v/v) and intravenously infused into the antecubital vein at a dose of 3 mg/kg with an infusion speed of 0.07 mL/s.
  Interventions: Drug: domestic polysaccharide superparamagnetic iron oxide nanoparticle

INTERVENTIONS:
Drug: domestic polysaccharide superparamagnetic iron oxide nanoparticle — Patients will receive contrast-enhanced renal magnetic resonance imaging with polysaccharide superparamagnetic iron oxide nanoparticle before renal angiography. Patients received intravenous polysaccharide superparamagnetic iron oxide nanoparticle before magnetic resonance imaging.
  Other Names: ferumoxytol

SUMMARY:
Conventional contrast-enhanced magnetic resonance imaging is typically performed with extracellular gadolinium chelates, which is often limited in patients with CKD owing to the risk of nephrogenic systemic fibrosis. Ferumoxytol, a novel contrast medium, can be used as an "off-label" contrast agent for magnetic resonance imaging. During the last decade, ferumoxytol has gained appeal as an MRI contrast agent in patients with estimated glomerular filtration rates <30mL/min and there are reports in the literature for its safe use and utility in both adult and pediatric patients with CKD. The study is designed to evaluate the diagnostic performance of ferumoxytol-enhanced magnetic resonance imaging in patients suspected of renal artery stenosis, investigate the correlation between renal cortical T2*(T2*=1/R2*) and renal function, and develop an automatic algorithms for renal vessel segmentation.

DETAILED DESCRIPTION:
This study is a single-center, prospective, controlled and diagnostic clinical trial to evaluate renal vasculature and renal function with ferumoxytol-enhanced magnetic resonance imaging using domestic polysaccharide superparamagnetic iron oxide injection as the contrast agent. This study will enroll 40 patients with or without renal impairment that are expected to undergo renal artery angiography in China. The investigators will record the baseline data of patients after admission. Patients will receive enhanced renal magnetic resonance imaging with polysaccharide superparamagnetic iron oxide nanoparticle to assess renal vasculature and renal function. The related laboratory indices will be reviewed at 24-72 h after magnetic resonance imaging, and then patients will receive renal angiography. The indices will be reexamined at 1 month and 3 months after magnetic resonance imaging. In order to evaluate the safety of polysaccharide superparamagnetic iron oxide nanoparticle, patients will detect iron levels in peripheral and tissue before and after the examination. The results of MR imaging including image quality, degree of vascular stenosis, and quantitative T2* values of the renal cortex will be evaluated independently by two experienced radiologists. The degree of stenosis of the same vessels assessed by Quantitative Coronary Analysis (QCA) will be used for comparison with MR results. All clinical adverse events will be recorded by investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18 years, < 75 years;
* Patients who planned renal angiography (hypertension 、renal failure、atherosclerosis）;
* Patients with normal renal function or CKD stage 1-5(Patients diagnosed with CKD as defined in the KDIGO Clinical Practice Guidelines for the Evaluation and Management of Chronic Kidney Disease 2012 Edition);
* Patients themselves or authorized families to sign informed consent voluntarily.

Exclusion Criteria:

* Patients who were allergic to iodine contrast agent or had allergic history or allergic constitution to iron and dextran;
* Patients who can't accept magnetic resonance examination because of psychological ( such as Claustrophobia ) or physical reasons ( such as metal retention in the body );
* Malignancies or other comorbid conditions with life expectancy less than 1 year;
* Pregnant or lactating women;
* Hearing impaired persons;
* Cardiac function grade III-IV;
* Patients who were taking other iron agents orally or intravenously;
* Patients with hemosiderin deposition or hemochromatosis;
* Patients with acute coronary syndromes;
* Any other patients that researcher deems it's unsuitable to be admitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
the degree of renal artery stenosis | baseline and after intervention
  Degree of renal artery stenosis assessed by Magnetic Resonance Imaging and renal angiography
quantitative cortical T2* value | baseline and after intervention
  the quantitative T2* value of the renal cortex will be measured bilaterally at the upper and lower poles by drawing six equal-sized, non-overlapping operator-dependent regions of interest (ROI) to calculate average quantitative T2* values.
change of hemoglobin level | baseline,72 hours,30 days,3 months
  hemoglobin examination of patients before and after examination to evaluate anemia.
serum creatinine | baseline,72 hours,30 days,3 months
  serum creatinine examination of patients before and after examination to evaluate kidney function.
Urine routine | baseline,72 hours,30 days,3 months
  Urine routine examination of patients before and after examination to evaluate kidney function.
24-hour urine biochemistry | baseline,72 hours,30 days,3 months
  24-hour urine biochemistry examination of patients before and after examination to evaluate kidney function.
Retinol binding protein | baseline,72 hours,30 days,3 months
  Retinol binding protein examination of patients before and after examination to evaluate kidney function.
Neutrophil gelatinase-associated lipocalin | baseline,72 hours,30 days,3 months
  Neutrophil gelatinase-associated lipocalin examination of patients before and after examination to evaluate kidney function.
Serum iron | baseline,72 hours,30 days,3 months
  Determination of serum iron before and after MRA to evaluate the changes of iron content in peripheral blood.
Ferritin | baseline,72 hours,30 days,3 months
  Determination of serum ferritin before and after MRA to evaluate the changes of iron content in peripheral blood.
Transferrin | baseline,72 hours,30 days,3 months
  Determination of serum transferrin before and after MRA to evaluate the changes of iron content in peripheral blood.
serum cystatin C | baseline,72 hours,30 days,3 months
  Determination of serum cystatin C before and after examination to evaluate the changes of renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr,PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No